CLINICAL TRIAL: NCT07153601
Title: Comparison of the Effectiveness of Bolus Doses of Norepinephrine 4 mcg and Phenylephrine 50 mcg in Managing Hypotension After Spinal Anesthesia in Cesarean Section Patients
Brief Title: Norepinephrine vs. Phenylephrine for Spinal Hypotension in Cesarean Section
Acronym: Norepinephrine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Imam Syahputra, dr, Universitas Sumatera Utara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 103/KEPK/USU/2025
Record Dates: First submitted 2025-07-08; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hypotenstion; Cesarean Resection; Anesthesia Spinal; Pregnancy Complications; Cardiovascular
MeSH Terms: conditions — Pregnancy Complications | interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norepinephrine Group (Experimental): Participants in this group received intravenous bolus doses of norepinephrine 4 mcg (2 mL) diluted in normal saline to treat spinal anesthesia-induced hypotension during cesarean section.
  Interventions: Drug: Norepinephrine 4mcg
- Phenylephrine Group (Experimental): Participants in this group received intravenous bolus doses of phenylephrine 50 mcg (2 mL) diluted in normal saline to treat spinal anesthesia-induced hypotension during cesarean section
  Interventions: Drug: Phenylephrine 50 mcg

INTERVENTIONS:
Drug: Norepinephrine 4mcg — Norepinephrine 4 mcg IV bolus diluted in 2 mL normal saline, administered upon onset of hypotension during spinal anesthesia.
  Arms: Norepinephrine Group
Drug: Phenylephrine 50 mcg — Phenylephrine 50 mcg IV bolus diluted in 2 mL normal saline, administered upon onset of hypotension during spinal anesthesia.
  Arms: Phenylephrine Group

SUMMARY:
This clinical trial was conducted to compare the effectiveness and safety of two medications-norepinephrine and phenylephrine-in treating low blood pressure (hypotension) that often occurs during spinal anesthesia for cesarean section (C-section) deliveries. Spinal anesthesia is commonly used during C-sections but can cause a drop in the mother's blood pressure, which may affect both the mother and the baby.

In this study, 46 pregnant women undergoing elective C-sections were randomly given either norepinephrine (4 mcg) or phenylephrine (50 mcg) when their blood pressure dropped. Researchers monitored their heart rate, blood pressure, and any side effects for 30 minutes after anesthesia.

The results showed that both drugs were effective in raising blood pressure. However, norepinephrine kept the heart rate more stable, while phenylephrine caused a noticeable slowing of the heart rate (bradycardia). Both drugs were safe and well tolerated.

This study suggests that norepinephrine may be a better option for managing low blood pressure during spinal anesthesia in C-sections, especially when maintaining heart rate and cardiac output is important.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-40 years
* Undergoing elective cesarean section
* Receiving spinal anesthesia
* Classified as ASA Physical Status II
* Stable baseline hemodynamics prior to anesthesia
* Not using inotropic, chronotropic, or vasoactive drugs before surgery

Exclusion Criteria:

* Emergency cesarean section
* Fetal distress
* Preeclampsia or eclampsia
* Contraindications to spinal anesthesia (e.g., coagulopathy, infection at injection site)
* Known allergy to norepinephrine or phenylephrine
* Hemodynamic instability prior to vasopressor administration
* Withdrawal from study or refusal to participate
* Failure to develop post-spinal hypotension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure (SBP) After Vasopressor Administration | Baseline to 2 minutes post-administration (T0-T2)
  Change in systolic blood pressure measured before vasopressor administration (T0-T1) and two minutes after administration (T2) in response to intravenous bolus of norepinephrine 4 mcg or phenylephrine 50 mcg during spinal anesthesia-induced hypotension in cesarean section patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Adam Malik Hospital, Medan, North Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-08-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT07153601/Prot_000.pdf